CLINICAL TRIAL: NCT04634435
Title: A Phase 1 Study of Autologous Memory-like Natural Killer (NK) Cell Immunotherapy With BHV-1100 and IVIG Followed by Low Dose IL-2 as Early Post-Autologous Transplant Consolidation in Minimal Residual Disease Positive, Multiple Myeloma (MM) Patients in First or Second Remission
Brief Title: Autologous Memory-like NK Cell Therapy With BHV-1100 and Low Dose IL-2 in Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BHV1100-101
Record Dates: First submitted 2020-10-21; First posted 2020-11-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Cell Therapy; CIML NK cell therapy; cytokine induced memory-like natural killer cell therapy; immunotherapy; antibody-dependent cell-mediated cytotoxicity; ADCC; CD38 positive; CD38+; plasma cells; multiple myeloma; hematological malignancies
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms | interventions — Immunoglobulins, Intravenous; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BHV-1100 Combination Treatment (Experimental)
  Interventions: Combination Product: BHV-1100 plus cytokine induced memory-like (CIML) NK cells plus IVIG and low dose IL-2

INTERVENTIONS:
Combination Product: BHV-1100 plus cytokine induced memory-like (CIML) NK cells plus IVIG and low dose IL-2 — Single dose infusion of BHV-1100 plus CIML NK Cells plus IVIG, followed by low dose IL-2

SUMMARY:
This is an open-label single center Phase 1a/1b study with the primary objective of establishing the safety and exploring the efficacy of infusing the ex vivo combination product of BHV-1100 plus cytokine induced memory-like (CIML) NK cells plus IVIG and low dose IL-2 in the peri-transplant setting in MM patients with minimal residual disease (MRD+) in first or second remission.

ELIGIBILITY:
Inclusion Criteria:

* Had measurable disease according to Standard Diagnostic Criteria at the time of initial Multiple Myeloma diagnosis
* Meets criteria for symptomatic multiple myeloma at the time of induction chemotherapy
* Is transplant eligible based on clinician judgement
* Willing to undergo ASCT in first or second remission
* Achieve partial response or better with induction chemotherapy prior to ASCT according to the IMWG Uniform Response Criteria for Multiple Myeloma
* Be MRD+ upon restaging prior to stem cell collection and ASCT
* Eastern Cooperative Oncology Group (EGOG) performance status score of less than 2
* Life expectancy greater than six months
* Have a creatinine clearance > 45 mL/min/m2 at the time of transplant evaluation
* If frozen stem cells from earlier mobilized leukapheresis are unavailable at the time of mobilized leukapheresis, patients must meet parameters/criteria according to institutional SOP for autologous stem cell apheresis
* Be willing and clinically stable to undergo stem-cell mobilized and collect enough CD34+ cells sufficient for 2 ASCT per institutional guidelines or investigator discretion or have sufficient frozen cells from a SoC collection prior to signing study consent
* Be willing and clinically stable to undergo a non-mobilized MNC-Apheresis while admitted to the hospital to generate CIML NK cells
* Be willing to undergo maintenance after ASCT per NCCN guidelines based on disease risk
* If a woman of child-bearing potential, be willing to follow birth control and pregnancy testing practice as recommended
* Be willing to undergo bone marrow aspirate and biopsy as per treatment plan
* Patients must meet adequate organ function/reserve based on institutional SOP for autologous stem cell transplant eligibility
* Non-secretory MM can participate if they have measurable disease in the bone marrow and are amenable to be followed by MRD testing

Exclusion Criteria:

* Prior autologous or allogeneic hematopoietic stem cell transplant
* Prior cellular therapies, including NK cell therapy
* Prior treatment with monoclonal antibodies, within 28 days of MCN apheresis
* Prior treatment with high dose melphalan
* Prior treatment with immunosuppressive or immunomodulatory agents with exception of 5 mg or less of prednisone daily, within 14 days of MCN-Apheresis
* Disease progression at the time of study treatment
* History of Plasma Cell Leukemia at any time prior to enrollment
* Patients seropositive for the human immunodeficiency virus (HIV)
* Uncontrolled, Hepatitis C Virus or Hepatitis B Virus infection
* Patient receiving other investigational therapy
* Patients with active, clinically significant autoimmune diseases
* Patients with active, clinically significant cancer other than multiple myeloma
* Patients with severe, uncontrolled psychiatric or neurological conditions that make difficult the assessment of neurologic toxicity of the study treatment
* Patients who have received anti-MM therapy (with the exclusion of monoclonal antibodies) within 14 days of study treatment
* More than two prior lines of anti-myeloma therapy, with induction therapy followed by maintenance being considered as one line and CyBorD to RVD transition in the absence of progressive disease being considered as one line

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities following Combination Product administration | 90-100 days post Combination Product administration
Incidence and severity of side effects related to the Combination Product | 90-100 days post Combination Product administration

SECONDARY OUTCOMES:
Rate of MRD (by ClonoSEQ®) conversion from positive to negative at 90-100 days after transplantation | 90-100 days post-ASCT
Rate of MRD conversion from positive to negative | 1 year post-ASCT
Rate of MRD conversion from positive to negative at any time during the maintenance phase | Start of maintenance therapy 90-100 days post ASCT until disease progression (approximately 2-3 years)
Rate of PFS | 1 year post Combination Product administration
Rate of OS | 1 year post Combination Product administration
Best overall response rate per the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma | 90-100 days post-ASCT, 1 year post-ASCT, and overall during maintenance phase (approximately 3 years)
Incidence and severity of cytokine release syndrome per ASBMT consensus grading | 100 days post Combination Product administration
Incidence and severity of other Immune-related toxicities by CTCAE version 5.0 | 100 days post Combination Product administration
PK of BHV-1100 by determining plasma Tmax | 4 days post Combination Product administration
PK of BHV-1100 by determining plasma Cmax | 4 days post Combination Product administration
PK of BHV-1100 by determining plasma Cmin | 4 days post Combination Product administration
PK of BHV-1100 by determining plasma AUC | 4 days post Combination Product administration
PK of BHV-1100 by determining plasma t1/2 | 4 days post Combination Product administration

CONTACTS AND LOCATIONS:
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No